CLINICAL TRIAL: NCT05832177
Title: Outreach Core Activities
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-22345; U54CA163068 (NIH)
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer Education; Spanish Language Cancer Education
MeSH Terms: interventions — Protein Biosynthesis; Residence Characteristics; Lunch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Community Members who attend Cancer CientoUno (101) program: Community members who opt to participate in the online Cancer CientoUno (101) training program. They will be asked to complete a registration survey and the programs self-paced educational modules. At the start of the course, they will be asked to complete a brief survey. After every module, they will be asked to complete a brief survey. In addition, community members will be asked to complete a midterm survey and a 6-month follow up survey.
  Interventions: Behavioral: Cancer CientoUno (101) program
- Community Members who Attend Symposium: Community members who opt to attend this symposium which will offer educational presentations focused on prevention, nutrition, clinical trials, and specific cancer types addressed in breakout sessions. Participants will be asked to complete a registration form and a post-event evaluation form.
  Interventions: Behavioral: Latinos y el cáncer/Hablemos de cáncer (Translation in English: Latinos and Cancer/Let's Talk About Cancer)
- Community Members who Attend Charlas (Talks): Community members who opt to attend these charlas (talks) which will offer education on a variety of cancer-related topics. The topics are selected in response to each event, given the community interest or need for a specific cancer-related topic. Participants will be asked to complete a registration form and a post-event evaluation form.
  Interventions: Behavioral: ¡Salud! Serie de Charlas (Translation in English: Health! Talk Series)
- Community Members who Attend Presentations: Community members who opt to attend and researchers (including those from the PHSU-MCC U54 partnership) will participate in these presentations to generate a discussion about ongoing research and have an opportunity for community members learn and provide feedback on on-going and completed research projects. Presentations from El Puente events will occur in Spanish (in Puerto Rico and Florida) and in English (in Florida). Attendees will be asked to complete a registration form and a post-event evaluation.
  Interventions: Behavioral: Community/Researcher Forum: El Puente (Translation in English: The Bridge).
- Community Members who Access Series of Virtual Lunch and Learn Podcasts: Community members will have access to a series of virtual Lunch and Learn podcasts, which will be 30-minute long, pre-recorded sessions in English and/or Spanish. Podcast sessions will cover updated cancer-relevant recommendations from the United States Preventive Services Task Force (USPSTF). Reach will be tracked with number of visits and/or other access metrics.
  Interventions: Behavioral: Lunch and Learn Updated Recommendations Series.
- U54 Partnership Investigators: These CE workshops will be mandatory for all partnership researchers who receive U54 funding in the proposed renewal period including Full, Pilot, and Developmental projects. The CE workshops are aimed to increase researchers' knowledge about the best strategies to establish teamwork with community members to achieve mutual benefits and advance translational research in cancer.
  Interventions: Behavioral: Community Engagement (CE) Training Program for U54 Partnership Investigators
- Lay Community Members: Lay community members will opt to participate in a 2-day CE workshop series. The goal is to include trained lay community members to actively participate in cancer prevention education and research. These activities will facilitate community-academic partnerships between the Partnership researchers and community members.
  Interventions: Behavioral: Community Engagement (CE) Training Program for Lay Community Members
- Community Members who Join Community Advisory Panel (CAP): The Community Advisory Panel (CAP) members will include individuals who are cancer survivors, family members/caregivers of cancer survivors, and/or representatives from healthcare, community- and faith-based organizations who are invited to join the CAP and accept the invitation. The PHSU-MCC Partnership utilizes a CAP to inform and guide overall outreach activities in PR and FL. Two CAPs, one at MCC and one at PHSU have been organized. Previous CAP members will be retained if interested and new CAP members added as needed.
  Interventions: Behavioral: Community Advisory Panels (CAP)
- U54 Partnership Investigators and CAP Members: During standing CAP meetings, partnership investigators present their ongoing research to members of the CAPs. Researchers who receive U54 funding in the proposed renewal period including Full, Pilot, and Developmental projects can request CAP feedback on topics along the research continuum from concepts for new research projects, ideas for recruitment, or dissemination of fundings.
  Interventions: Behavioral: Research Corner
- Community Leaders and Stakeholders: Community leaders from disadvantaged socioeconomic areas and Stakeholders of healthcare organizations with whom the Program has established previous collaborative relationships will participate in the CBTP. The stakeholders include nurses, community health educators, clinical social workers, among other healthcare professionals.
  Interventions: Behavioral: Community-based Training Program (CBTP) for Community Leaders and Stakeholders.
- Stakeholders: Physicians, nurses, psychologists, and other stakeholders within the communities under the partnership umbrella will participate in the Cancer 101 Stakeholders program.
  Interventions: Behavioral: Integrate Cancer 101 into the Stakeholders Programs

INTERVENTIONS:
Behavioral: Cancer CientoUno (101) program — The Spanish version of Cancer 101 consists of several modules that address cancer control and prevention, risk factors, early detection and screening guidelines, cancer diagnosis and stages, cancer treatment, cancer and genetics, cancer and chronic disease, patient and caregiver support, HPV, biobanking, and clinical trials. All modules contain a written summary with learning objectives, a PowerPoint presentation, pre- and post-module evaluations with an answer sheet, a glossary, references, and supplemental resources. This program will occur on an ongoing basis.
  Groups: Community Members who attend Cancer CientoUno (101) program
Behavioral: Latinos y el cáncer/Hablemos de cáncer (Translation in English: Latinos and Cancer/Let's Talk About Cancer) — This is a biennial cancer symposium focused on cancer topics important to Hispanic/Latinos. This day-long event includes a plenary session and concurrent sessions where healthcare professionals present educational information about cancer, cancer prevention, early detection methods, and other related topics.
  Groups: Community Members who Attend Symposium
Behavioral: ¡Salud! Serie de Charlas (Translation in English: Health! Talk Series) — This is an educational and community outreach effort comprised of local charlas (talks) led by Hispanic/Latino healthcare professionals (e.g., the partnership Community Health Educator [CHE], topic experts) who provide education and answer questions about specific cancer topics. The charlas may be conducted in multiple modalities (in person, virtual, hybrid) and may be conducted in English and/or Spanish. At least three events will be held each year in the partnership locations.
  Groups: Community Members who Attend Charlas (Talks)
Behavioral: Community/Researcher Forum: El Puente (Translation in English: The Bridge). — The main goal of the El Puente annual event is to generate dialogue between community members and researchers about cancer treatment and cancer-focused research topics. During El Puente's presentations, researchers present their projects and data results to community members, allowing community members to react to the research, make suggestions, and express concerns.
  Groups: Community Members who Attend Presentations
Behavioral: Lunch and Learn Updated Recommendations Series. — This is a virtual podcast that will discuss cancer-related recommendations and guidelines from the United States Preventive Services Task Force (USPSTF). The podcasts are pre-recorded, 30 minute long, and will be in English and/or Spanish. This podcast will be hosted by the Outreach Core (OC) CHE, and feature experts who will explain the updated recommendations and active steps that community members and providers can take to facilitate adherence. This activity will begin according to the project timeline
  Groups: Community Members who Access Series of Virtual Lunch and Learn Podcasts
Behavioral: Community Engagement (CE) Training Program for U54 Partnership Investigators — This is a series of 2 1/2-day CE workshops designed and delivered up to 20 partnership researchers (including faculty and junior investigators) delivered across four sessions per year (6 to 10 researchers per year). Each session includes two hours of lectures (didactic material) and one hour of practice activities (practical application of the theoretical content). Session topics will include CE: concepts and principles, theoretical roots, levels, and ethics. The OC team will provide educational materials and additional references in each session.
  Groups: U54 Partnership Investigators
Behavioral: Community Advisory Panels (CAP) — These CAPs work closely with the (CHE) to oversee the identification, development, and coordination of the outreach activities; provide advice on the development and implementation of community needs and assessments; provide guidance for recruitment and retention of research participants; and assist in the recruitment for educational events and research and vetting community educational materials and the content of protocols for research projects.
  Groups: Community Members who Join Community Advisory Panel (CAP)
Behavioral: Research Corner — The goal is to provide bidirectional communication between the community and researchers to increase CE strategies into cancer disparities research through periodic meetings between community members and researchers to discuss CE strategies, research recruitment strategies, dissemination strategies, among others.
  Groups: U54 Partnership Investigators and CAP Members
Behavioral: Community-based Training Program (CBTP) for Community Leaders and Stakeholders. — The CBTP provides the opportunity to acquire knowledge to impart cancer prevention education (Cancer 101) and skills necessary to disseminate educational information (hands-on experiences through OC educational activities). This training will be provided in-person and remotely to increase participation. This activity will begin according to the project timeline.
  Groups: Community Leaders and Stakeholders
Behavioral: Integrate Cancer 101 into the Stakeholders Programs — This program will offer stakeholders a no-cost workshop of three credit hours to increase cancer prevention education among Hispanic/Latinos. CMEs will be provided virtually to increase participation. This activity will begin according to the project timeline.
  Groups: Stakeholders
Behavioral: Community Engagement (CE) Training Program for Lay Community Members — A series of two-day CE workshops designed and delivered to 30 lay community members over a four-year period (6 to 10 participants per year). The proposed CE workshops includes: 1) CE principles, 2) cancer prevention education principles, and 3) community-based promotion strategies for cancer prevention. This activity will begin according to the project timeline.
  Groups: Lay Community Members

SUMMARY:
The Outreach Core (OC) of the Ponce Health Sciences University-Moffitt Cancer Center (PHSU-MCC) Partnership provides community outreach and education to improve cancer screening behaviors in our catchment area populations. The overall goal of the OC is to increase community cancer awareness, community engagement, and participation in cancer research and outreach in our catchment areas. Working closely with other Partnership cores and investigators, the team proposes to elevate and expand its activities to facilitate reciprocal communication between community members and partnership researchers through OC educational activities, training opportunities, supporting participant recruitment efforts, and incorporating the Community Advisory Panel (CAP) feedback on partnership research projects. Together with community members and Partnership researchers, the OC will increase cancer awareness, community engagement, and participation in cancer research in communities served by MCC (in FL) and PHSU (in PR) through the following three Specific Aims:

Aim 1: To develop, deliver, and disseminate cancer education and outreach activities to our catchment area populations. The team will deliver cancer education to communities in PR and FL using evidence-based programs through multiple delivery strategies and reflecting partnership research priorities and topics of interest identified by community members.

Aim 2: To enhance capacity for mutually beneficial research engagement to address cancer health priorities in our catchment areas. The team will facilitate communication between community members and partnership investigators (e.g., CAP Research Corner), support partnership research that is responsive to community needs (translational research), promote community participation in the partnership's research activities/projects, and train researchers and community members in community engagement principles.

Aim 3: To expand the capacity to train community members as lay health promoters to deliver evidence-based cancer education programs in their communities. The team will train community members and community partners/organizations to deliver evidence-based cancer education (e.g., Cancer 101, OC activities) in their local communities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Any health status
* Able to speak, read and write Spanish or English (some events are in Spanish, some are in English)
* [Cancer 101 Online Training Program, Lunch and Learn podcast, and Stakeholders Program only]: Have access to the internet
* Willing to complete the training modules and assessments [Cancer 101 Online Training Program]
* Willing to complete registration, attendance logs, and evaluations, as applicable
* [Community Engagement Training Program, Research Corner only]: be a researcher who received U54 funding in the proposed renewal period including Full, Pilot, and Developmental projects.
* [Stakeholders in the Community-based Training Program and Cancer 101 Stakeholders program only]: nurses, community health educators, clinical social workers, physicians, psychologists, among other healthcare professionals

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community members who are physicians, nurses, psychologists, community health educators, and clinical social workers
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants that Complete the Cancer 101 Online Training Program | At 15 Weeks from Start of Training Program
  Program completion data will be based upon whether individuals complete the modules and assessments
Number of Participants that Access the Cancer 101 Online Training Information Post Training | At 6 months Post Training Program
  Number of participants that access the online program after completing the online training program
Changes in cancer-related knowledge and self-efficacy for providing health education | Day 1 and upon completion of Cancer 101 Online Training program, 15 weeks
  Data will be based on self-reported assessments completed by Cancer 101 online program participants prior to starting the course and upon completion of the course
Number of participants that attend Latinos y el cáncer/Hablemos de cáncer symposia | Day 1
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of participants that attend ¡Salud! Serie de Charlas events | Day 1
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of participants that attend El Puente events | Day 1
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of participants that access recordings of the Lunch and Learn podcast | 1 week after posting, 1 month after posting, 6 months after posting
  Data will be based on event tracking related to access to podcast recordings
Number of U54 partnership investigator participants that attend the Community Engagement (CE) Training Program | Day 1 and Day 3, at start of and upon completion of each Community Engagement Training Program workshop]
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of community member participants that attend the Community Engagement (CE) Training Program | Day 1 and Day 2 of at start and upon completion of each Community Engagement Training Program]
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of CAP meetings held per year and number of CAP members | Day 1
  Data will be based on event tracking metrics for attendance
Number of Research Corner presentations presented at CAP meetings | Day 1
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of trainees that complete the Community-based Training Program (CBTP) for Community Leaders and Stakeholders | Day 1 and Day 3, at start of and upon completion of the Community-based Training Program)
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of trainees that complete the Cancer 101 Stakeholders Program | Upon completion of the Stakeholders Program, 15 weeks
  Data will be based on event tracking metrics for attendance and evaluation completion
Number of Cancer 101 Stakeholders Program trainees that complete CME credits | Upon completion of the Stakeholders Program, 15 weeks
  Data will be based on event tracking metrics for CME completion

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Christy, PhD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- Moffitt Cancer Center, Tampa, Florida, United States
- Ponce Health Sciences University, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=22345